CLINICAL TRIAL: NCT07356245
Title: Phase II Study of Ruxolitinib Maintenance Post-Hematopoietic Stem Cell Transplant in T-Cell Lymphoma
Brief Title: Ruxolitinib Maintenance Post-Hematopoietic Stem Cell Transplant T-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonathan Brammer (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Brammer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24353; NCI-2026-00140 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2026-01-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: T-cell Lymphoma; Graft Versus Host Disease; Lymphoma, T-Cell; Peripheral T Cell Lymphoma; T-cell Prolymphocytic Leukemia; Cutaneous T Cell Lymphoma; Adult T-cell Leukemia/Lymphoma; Primary Cutaneous T-Cell Non-Hodgkin Lymphoma
Keywords: stem cell transplant; graft versus host disease; lymphoma; leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Graft vs Host Disease; Lymphoma, T-Cell, Peripheral; Leukemia, Prolymphocytic, T-Cell; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Leukemia | interventions — ruxolitinib; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib maintenance) (Experimental): Starting day +35 to day +120 post-SCT, patients receive ruxolitinib PO BID on days 1-30 of each cycle. Cycles repeat every 30 days for 1 year post-SCT, in the absence of disease progression or unacceptable toxicity. Patients undergo PET-CT scan and blood sample collection throughout the study. Patients may undergo bone marrow biopsy and/or tissue biopsy throughout the study, at time of progression.
  Interventions: Drug: Ruxolitinib; Procedure: Positron emission tomography-computed tomography; Procedure: Bone Marrow Biopsy; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Ruxolitinib — Administered orally twice daily
Procedure: Positron emission tomography-computed tomography — Undergo PET-CT Scan
  Other Names: PET-CT; PET-CT Scan; Computed tomography
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological sampe collection; Biospecimen Collected; Speciment collection

SUMMARY:
This phase II trial tests how well ruxolitinib as a maintenance medication works to prevent relapse and graft-versus-host disease (GVHD) for patients who have undergone stem cell transplantation for T-cell lymphoma. GVHD is a common problem that may occur after a blood stem cell transplant. The "graft" is the donor blood cells that patients get during the transplant. The "host" is the person receiving the cells. GVHD is when the donor graft attacks and damages some of the transplant recipient's tissues. Ruxolitinib is a type of drug called a Janus kinase (JAK) inhibitor which works by decreasing the immune response of cells in the body. It is also a cancer growth blocker that blocks the growth factors that trigger the cancer cells to divide and grow. Ruxolitinib works by blocking a gene, called JAK2, that is important in the production of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of ruxolitinib phosphate (ruxolitinib) on relapse at 1-year after autologous (auto) stem cell transplant (SCT) in T-cell lymphoma (TCL).

II. Determine the effect of ruxolitinib on graft versus host disease (GvHD) and relapse free-survival (GRFS) at 1-year for allogeneic (allo) SCT in TCL.

SECONDARY OBJECTIVES:

PRIMARY OBJECTIVES:

I. Determine the effect of ruxolitinib phosphate (ruxolitinib) on relapse at 1-year after autologous (auto) stem cell transplant (SCT) in T-cell lymphoma (TCL).

II. Determine the effect of ruxolitinib on graft versus host disease (GvHD) and relapse free-survival (GRFS) at 1-year for allogeneic (allo) SCT in TCL.

SECONDARY OBJECTIVES:

I. Survival (progression free survival [PFS]/overall survival [OS]) of patients with ruxolitinib maintenance (auto-SCT, allo-SCT, whole cohort).

II. Determine the safety and feasibility of ruxolitinib maintenance post-SCT. III. Determine the effect of ruxolitinib on the cumulative incidence (CI) of grade II-IV acute GVHD (alloSCT), chronic extensive GVHD, non-relapse mortality (NRM) (auto-SCT and allo-SCT).

EXPLORATORY OBJECTIVES:

I. Determine the effect of maintenance ruxolitinib compared to matched historical controls using the Center for International Blood and Marrow Transplant Research (CIBMTR) registry.

II. Determine the effect of ruxolitinib on immune modulation and reconstitution post-allo-SCT and upon disease relapse.

OUTLINE:

Starting day +35 to day +120 post-SCT, patients receive ruxolitinib orally (PO) twice daily (BID) on days 1-30 of each cycle. Cycles repeat every 30 days for 1 year post-SCT, in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET)-computed tomography (CT) scan and blood sample collection throughout the study. Patients may undergo bone marrow biopsy and/or tissue biopsy throughout the study, at time of progression.

After completion of study treatment, patients are followed up at 18 and 24 months then yearly until 5 years and at progression.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with T-cell lymphoma [PTCL (all subtypes), T-PLL, ATLL, and CTCL (all subtypes)] in partial or complete remission between day +35 and +120 from auto-SCT or allo-SCT
2. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
3. Adequate hematologic function defined by absolute neutrophil count (ANC) > 1000/mm3 without granulocyte colony-stimulating factor (G-CSF) for at least 3 days, platelets > 50K/mm3 without transfusion for at least 3 days and hemoglobin (Hb) > 8.0 g/dL without transfusion for at least 3 days.
4. Adequate organ function defined by total Bilirubin < 1.5 x ULN, alanine aminotransferase (ALT) </= 3 x ULN, CKD-EPI eGFR ≥ 30 ml/min, SpO2 > 92% without supplemental oxygen and ejection fraction more than 45%.
5. Able to tolerate oral or enteral medications.
6. Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.
7. Able to read and sign informed consent.

Exclusion Criteria:

1. Anaplastic lymphoma kinase (ALK)+ or Dual specificity 22 (DUSP22)+ ALCL with low international prognostic index (IPI) score (<2) in first complete remission.
2. Progressive disease or any other systemic therapy post-SCT (radiation allowed)
3. Disease progression to Ruxolitinib previously
4. GvHD requiring systemic therapy.
5. Active uncontrolled infections.
6. Active thrombotic active microangiopathy requiring therapy.
7. History of veno-occlusive disorder post-transplant
8. Use of platelets antiaggregant or anticoagulants deemed to be unsafe to be held in case of thrombocytopenia.
9. History of life-threatening bleeding defined as any bleeding that required invasive procedures or involving central nervous system.
10. Pregnancy (positive Beta HCG test in a woman with childbearing potential defined as not postmenopausal for 12 months or no previous surgical sterilization) or currently breast-feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
11. Uncontrolled Hepatitis B/C, HIV, tuberculosis, mycobacterium, or fungal infection.
12. Exposure to other investigational drugs within 4 weeks before enrollment.
13. Grade ≥ 3 non-hematologic toxicity from SCT that has not resolved to grade ≤ 2.
14. Myocardial infarction or stroke within 1 year of study entry.
15. Any uncontrolled medical problem at the discretion of the investigator that would pose a risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence (CI) of relapse | at 1-year post-auto-SCT
  Relapse is defined as evidence of disease progression or recurrence based on Lugano criteria or confirmed by biopsy.
GvHD and relapse free-survival (GRFS) | at 1-year post-allo-SCT
  GRFS is a composite endpoint of survival without grade III-IV acute GVHD, systemic therapy-requiring chronic GVHD (cGVHD), relapse, or death. Will be evaluated using the Kaplan-Meier method, with median survival and probability of surviving to relevant time points reported with point estimates and 90% confidence intervals separately for each study cohort. Comparisons to Center for International Blood and Marrow Transplant Research (CIBMTR) patients will use log-rank tests.

SECONDARY OUTCOMES:
Progression-Free survival (PFS) | At 1 and 2 years
  Will be evaluated using the Kaplan-Meier method, with median survival and probability of surviving to relevant time points reported with point estimates and 90% confidence intervals separately for each study cohort. Comparisons to CIBMTR patients will use log-rank tests
Overall Survival (OS) | At 1 and 2 years
  Will be evaluated using the Kaplan-Meier method, with median survival and probability of surviving to relevant time points reported with point estimates and 90% confidence intervals separately for each study cohort. Comparisons to CIBMTR patients will use log-rank tests.
Cumulative incidence of grade II-IV acute GVHD (allo-SCT cohort) | Up to 5 years
  Will be conducted using non-relapse mortality (NRM) as a competing risk, with estimates of cumulative incidence at various time points reported with 90% confidence intervals. Cumulative incidences will be compared to CIBMTR data using Fine-Gray analysis.
Cumulative incidence of chronic extensive GvHD (allo-SCT cohort) | at 1 year post-SCT
  Will be conducted using NRM as a competing risk, with estimates of cumulative incidence at various time points reported with 90% confidence intervals. Cumulative incidences will be compared to CIBMTR data using Fine-Gray analysis.
Cumulative Incidence of non-relapse mortality (NRM) at 1-year after (auto-SCT, allo-SCT, whole cohort) | At 1 year
  Will be conducted using NRM as a competing risk, with estimates of cumulative incidence at various time points reported with 90% confidence intervals. Cumulative incidences will be compared to CIBMTR data using Fine-Gray analysis
Rates of grade 3-4 treatment Emergent Adverse Events | Up to 2 years
  Treatment-emergent adverse events of grade 3 and higher will also be reported for each cohort
Rate of patients completing 1-year post-SCT maintenance Ruxolitinib | At 1 year post-SCT
  Will be conducted using NRM as a competing risk, with estimates of cumulative incidence at various time points reported with 90% confidence intervals. Cumulative incidences will be compared to CIBMTR data using Fine-Gray analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Brammer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu